CLINICAL TRIAL: NCT02194413
Title: Effects of Healing Touch on Patients Undergoing Hematopoietic Stem Cell Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Susan Lutgendorf, Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201111724; P30CA086862 (NIH)
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Anxiety Disorder; Fatigue; Hematopoietic/Lymphoid Cancer; Pain
MeSH Terms: conditions — Anxiety Disorders; Fatigue; Hematologic Neoplasms; Pain | interventions — Therapeutic Touch; Touch

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (healing touch) (Experimental): Patients receive daily HT sessions comprising pain drain, chakra connection, magnetic clearing, and mind clearing over 30 minutes from day 1 until 2 days before discharge from the hospital (therapeutic touch).
  Interventions: therapeutic touch, quality-of-life assessment, and questionnaire administration
  Interventions: Procedure: therapeutic touch; Other: quality-of-life assessment; Other: questionnaire administration
- Arm II (usual care) (Active Comparator): Patients receive routine nursing care from doctors and nurses from day 1 until 2 days before discharge from the hospital.
  Interventions: quality-of-life assessment, and questionnaire administration
  Interventions: Other: quality-of-life assessment; Other: questionnaire administration

INTERVENTIONS:
Procedure: therapeutic touch — receiving healing touch
  Other Names: healing touch
  Arms: Arm 1 (healing touch)
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: questionnaire administration — Ancillary studies

SUMMARY:
This randomized pilot clinical trial studies healing touch or usual care in improving quality of life in patients undergoing stem cell transplant. Healing touch may improve the quality of life of patients undergoing stem cell transplant.

DETAILED DESCRIPTION:
Primary Objectives:

I. To estimate the effects of healing touch (HT) vs usual care in the following clinical outcomes of stem cell transplant (SCT) patients; length of hospital stay, days to engraftment, and number of hospital readmissions during 100 days post-transplant.

II. To estimate changes in quality of life (QoL) which occur during hospitalization of SCT patients who receive HT vs. usual care.

III. To examine differences in effects of HT vs. usual care (UC) in patients receiving related allogeneic (Allo) transplant compared to those receiving autologous (Auto) transplant.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive daily HT sessions comprising pain drain, chakra connection, magnetic clearing, and mind clearing over 30 minutes from day 1 until 2 days before discharge from the hospital.

ARM II: Patients receive routine nursing care from doctors and nurses from day 1 until 2 days before discharge from the hospital.

After completion of study treatment, patients are followed up for 100 days.

ELIGIBILITY:
Inclusion Criteria:

* Currently undergoing autologous (auto) or related allogeneic (related allo) stem cell transplantation
* Admitted to the University (U) Adult Blood and Bone Marrow Transplant Unit (UIBMTU) of the University of Iowa Hospitals and Clinic
* Ability to provide written informed consent obtained prior to participation in the study and able to complete questionnaires
* Pregnant woman who are eligible for stem cell transplant are included in this study

Exclusion Criteria:

* Patients with any significant history of non-compliance to medical regimens, with inability to grant a reliable informed consent or unable to complete questionnaires
* Patients with evidence of a significant psychiatric disorder by history that would prevent completion of the study will not be allowed to participate, i.e., schizophrenia, anxiety disorder, major depressive disorder and bipolar disorder
* Diagnosis of dementia or other disease affecting cognitive function
* Nursing women are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2017-01-18 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay, Days to engraftment defined as absolute neutrophil count (ANC: segs + bands) greater | Up to 100 days
Changes in QoL (POMS-SF, FACT-BMT, CES-D) | Baseline up to 100 days
  Changes in levels of QoL measures before and after hospitalization will be compared using the paired t-test or the nonparametric paired sign test, if the assumption of normality is substantially violated.

SECONDARY OUTCOMES:
Number of hospital readmissions | Up to 100 days

CONTACTS AND LOCATIONS:
Overall Officials: Susan K Lutgendorf, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No